CLINICAL TRIAL: NCT06082661
Title: Blood Collection for Use with Translational, Biomedical Research At UCF College of Medicine and Burnett School of Biomedical Sciences
Brief Title: Blood Collection for COM/BSBS
Status: Recruiting | Type: Observational
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00003409
Record Dates: First submitted 2023-10-03; First posted 2023-10-13 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: Blood; Healthy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this biospecimen collection protocol is the acquisition of blood from adult volunteers. These biospecimens will be transferred to the College of Medicine (COM)/Burnett School of Biomedical Sciences (BSBS) research scientists and their research teams for testing according to their separate IRB-approved/exempted protocols. These separate IRBapproved protocols cannot be for genetic testing.

DETAILED DESCRIPTION:
Research scientists of the University of Central Florida College of Medicine (COM) and Burnett School of Biomedical Sciences (BSBS) conduct laboratory studies in biomedical and translational research for the purpose of understanding human disease and developing innovative methods for diagnosing, measuring, or treating disease or disease symptoms. The key research divisions are cancer, cardiovascular, immunity and pathogenesis, neuroscience, and molecular microbiology. Frequently, these studies require human blood (or its derivatives) for testing of assays and devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* 18 years old or older
* weigh over 110 pounds
* able to provide informed consent

Exclusion Criteria:

* pregnant/suspect to be pregnant
* prisoners
* have donated blood anywhere in the preceding 16 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study does not specifically target a particular vulnerable population.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Acquisition of blood samples for testing | 5 years
  This is a non-clinical, biospecimen collection study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No